CLINICAL TRIAL: NCT04476745
Title: The Effect of Weekly 50,000 IU Vitamin D3 Supplements on the Serum Levels of Selected Cytokines Involved in Cytokine Storm of Covid-19; A Randomized Clinical Trial in the Covid-19 Uninfected Jordanian People With Vitamin D Deficiency
Brief Title: The Effect of D3 on Selected Cytokines Involved in Cytokine Storm in the Covid-19 Uninfected Jordanian People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Principal Investigator, Mahmoud Suleiman Abu-Samak, Mahmoud S Abu-Samak, PhD Study Principal Investigator Department of Clinical Pharmacy and Therapeutics, Applied Science Private University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-PHA-16
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Cytokine Storm
Keywords: Covid -19; uninfected; IL-1; IL-6; TNF; VDD; Vitamin D3; 50,000IU
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: VD3 group (Experimental): Dietary Supplement: Dietary Supplement: Vitamin D3 Dietary Supplement: Vitamin D3 (50,000) IU / week for 8 weeks Other Names: cholecalciferol,
  Interventions: Dietary Supplement: Vitamin D3
- Control group (No Intervention): Control group No intervention was given

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Dietary Supplement: Vitamin D3 (50,000) IU / week for 8 weeks
  Other Names: cholecalciferol
  Arms: Experimental: VD3 group

SUMMARY:
The effect of Weekly 50,000 IU vitamin D3 supplements on the serum levels of selected cytokines involved in cytokine storm of Covid-19; A randomized clinical trial in the Covid-19 uninfected people with vitamin D deficiency.

DETAILED DESCRIPTION:
No data are available on the effect of Weekly 50,000 IU vitamin D3 supplements on the serum levels of selected cytokines involved in cytokine storm of Covid-19 in the Covid-19 uninfected Jordanian people with vitamin D deficiency. This study was designed to investigate whether a high dose of vitamin D3 (50,000 IU) / week for 8 weeks supplementation has a potential effect on cytokine storm of Covid-19; such as IL-1 beta, IL-6, and TNF in the Covid-19 uninfected Jordanian people with vitamin D deficiency.

This study aims to assess whether high doses of vitamin D3 may improve immune responses against COVID-19 infection in uninfected Jordanian peoples. We hypothesize that Weekly 50,000 IU vitamin D3 supplements will significantly change immune responses compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

Age ≥30 years old Male and female Jordanian ASU students and employees who live in Amman. Informed written consent from the participant prior to the start of the study. a serum 25(OH)D concentration less than 30 ng/mL.

Exclusion Criteria:

Any eligible subject refuses to apply with informed written consent before the start of the study. Men or women previously diagnosed with chronic diseases, including kidney disease or GIT problems. Who are receiving vitamin D3 supplements (3 months before the start of the study). Pregnant, Breastfeeding females, Females using hormonal contraceptives

Ages: 30 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
IL-1 beta | 8 weeks
  seum levels
IL-6 | 8 weeks
  serum levels
TNF | 8 weeks
  serum levels

SECONDARY OUTCOMES:
serum concentrations of 25-hydroxyvitamin D | 8 weeks
  ng/ml

OTHER OUTCOMES:
lipid profile parameters | 8 weeks
  seum levels

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Study Chair — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan; Dana A Bader, MSc, Principal Investigator — Department of Clinical Pharmacy and Therapeutics , Applied Science Private University, Amman -Jordan
Locations (1):
- Mahmoud S Abu-Samak, Amman, Jordan